CLINICAL TRIAL: NCT04396392
Title: VR-based Training for Adolescents With Fear of Public Speaking, a Randomized Controlled Trial
Brief Title: VR-based Exposure Training for Adolescents With Fear of Public Speaking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 60628
Record Dates: First submitted 2020-02-11; First posted 2020-05-20 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Mental Health Issue; Adolescent Development; Technology

STUDY DESIGN:
Intervention Model Description: The study is a two-phased intervention study
  Participants with PSA will be randomized into three self-guided intervention groups and one delayed waiting list group as follows:
  Group 1: receiving VR intervention (3 weeks)
  Group 2: receiving VR intervention (3 weeks) + text-based exposure program (T-B-Exp) (3 weeks)
  Group 3: receiving text-based psychoeducation and exposure program (T-B PE + T-B Exp) (6 weeks)
  Group 4: Waitlist (3 weeks) + receiving text-based psychoeducation (T-B PE) (3 weeks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR-based training (Experimental): receiving only VR intervention
  Interventions: Behavioral: VR-based training
- text-based training (Active Comparator): receiving only text-based intervention
  Interventions: Behavioral: VR-based training
- VR- and text-based training (Experimental): receiving both VR intervention and text-based intervention
  Interventions: Behavioral: VR-based training
- waiting list (No Intervention): waiting list in phase 1 and text-based training after 3 weeks

INTERVENTIONS:
Behavioral: VR-based training — All interventions will be home-based and self-guided. The participants will work on the interventions after school hours at home.
  All participants will be randomized into four groups (see Figure 1). All participants will receive an introduction module, with information tailored to their study group. Parents will receive an introduction module with information about the study group their adolescents belong to.
  Other Names: text-based training
  Arms: VR- and text-based training; VR-based training; text-based training

SUMMARY:
Public speaking anxiety (PSA) is a common anxiety with onset in adolescence and early adulthood. With the advent of consumer Virtual Reality (VR) technology, VR-delivered exposure therapy has previously been shown to be efficacious with adults. Virtual reality has existed for several decades, but it is only in the recent years it has become readily available. The new generation of off-the-shelf, consumer VR hardware, can revolutionize the design, availability and dissemination of VR therapist tools for exposure therapies. Importantly, there has been relatively little research on VR delivered exposure of anxiety in social situations compared to other anxiety disorders, presumably due to the complexity of the virtual stimuli required. There has been no study on VR delivered exposure specifically for adolescents until recently. A feasibility and pilot trial laying the foundation of the current study showed great potential in using VR for adolescents with PSA. The current study aims to investigate the efficacy of a self-guided VR intervention compared to a self-guided internet-delivered text-based intervention using a two-phased randomized design. Adolescents aged 13-16 will be invited to participate in the study

DETAILED DESCRIPTION:
The study is a two-phased intervention study .

Participants with PSA will be randomized into three self-guided intervention groups and one delayed waiting list group as follows:

Group 1: receiving VR intervention (3 weeks)

Group 2: receiving VR intervention (3 weeks) + text-based exposure program (T-B-Exp) (3 weeks)

Group 3: receiving text-based psychoeducation and exposure program (T-B PE + T-B Exp) (6 weeks)

Group 4: Waitlist (3 weeks) + receiving text-based psychoeducation (T-B PE) (3 weeks)

Interventions:

1. The VR intervention is a self-guided and home-based VR intervention that lasts for three weeks and focuses on exposure training. The VR group will receive the VR headset personally, in addition to instructional text about how the VR intervention works, how to use the VR application and how often to train. They will be instructed at least 5 tasks weekly during the intervention program.
2. The text-based Psychoeducation intervention is a three weeks program with three modules. One module will be assigned weekly, together with the weekly assessments, which will be same for all participants. The participants will receive a notification on text message when a module has been assigned to them. Module 1 will include information about the intervention program, psychoeducation about public speaking anxiety, cognitive therapy and case formulation. Module 2 will focus on catastrophic beliefs; how to recognize, how they develop, how they contribute to maintaining the anxiety and how they can be tested. Module 3 focuses on safety strategies; what they are, how they contribute in maintaining anxiety, and how to identify them.
3. The Text-based exposure intervention is a three weeks program with 3 modules. One module will be assigned weekly, together with weekly assessments. The modules will focus on how to practice exposure in real life (in vivo) and relapse prevention.
4. The waitlist group will be in waitlist mode for three weeks while the intervention groups are in phase 1. They will still receive weekly assessments during phase 1.

ELIGIBILITY:
Inclusion Criteria: Inclusion:

Aged 13-16, Symptoms of PSA, as defined by Public Speaking Anxiety Scale (PSAS) which leads to distress and / or negative consequences at school. Based on data from the feasibility study (Kahlon et.al 2019) the cut-off will be PSAS < 55.

-

Exclusion Criteria:

Current ongoing treatment for mental health problems (psychoactive medication/psychotherapy) impaired eyesight and lack of stereoscopic vision which cause difficulties in the VR experience and balance problems

-

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-03 (Estimated); Study Completion 2022-03-03 (Estimated)

PRIMARY OUTCOMES:
Change in Public Speaking Anxiety Scale | 18 months
  A new, modern, reliable and valid self-rating scale (Bartholomay & Houlihan, 2016). The PSAS features 17 items (5 of which are reverse-coded) covering cognitive, behavioral and physiological aspects of PSA. Since the PSAS features a full Likert item response format, it should be more sensitive to change than older rating scales such as the Personal Report of Confidence as a Speaker (Phillips, Jones, Rieger, & Snell, 1997). Normative score data is however as of yet missing. This scale is translated into Norwegian according to scientific standards (back-translation.). Although intended for adults, the wording did not present any problem for adolescents in our feasibility study. lower score means lower symptom-leves

SECONDARY OUTCOMES:
Change in Social Interaction Anxiety Scale | 18 months
  Fear of social interaction distinguishes performance-only from generalized SAD. As such, degree of social interaction anxiety is a likely moderator of treatment response in the current study. A combination of Social Interaction Anxiety Scale (SIAS) 6 and the Social Phobia Scale (SPS) 6 has proven to be a validated measure to measure the more generalized form of social anxiety and gives us a short screening tool which is easy to assess (Peters, Sunderland, Andrews, Rapee, & Mattick, 2012). This scale is translated into Norwegian according to scientific standards (back-translation.).
  By collecting data on the 12-item short version of SIAS at both pre and post and FU the aim is to investigate whether VRET for PSA has a treatment effect on generalized social anxiety lower score means lower symptom-levels. scale from 0-80.
Change in Catastrophic belief expectancy | 18 months
  Expectancy ratings of aversive consequences are a valid, simple way of assessing the strength of conditioning (Boddez et al., 2013) and a hypothesis is that a decrease in catastrophic beliefs expectancies will also cause a reduction in PSA symptoms . One-item scale for CBE will be assessed weekly together with the primary outcome measure PSAS. They will be asked to answer, "How sure are you that the most aversive consequence when giving a speech is likely to happen?" on as scale from 0-100.
  Alternative: "How sure are that you will sweat, shake, and/or rødme visibly? How sure are you that you will speak in a weird way? (snakke rart). How sure are you that you will have difficulties speaking? How sure are you that others will think negatively of you?
Change in Social Phobia Scale | 18 months
  Fear of social performance, By collecting data on the 12-item short version of SPS at both pre and post and FU the aim is to investigate whether VRET for PSA has a treatment effect on performance social anxiety.
  lower score means lower symptom-levels. scale from 0-80.

CONTACTS AND LOCATIONS:
Locations (1):
- Bergen Municipality Division School, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Not decided how this should be done yet